CLINICAL TRIAL: NCT04649892
Title: Predicting Response to Naltrexone With Eye Tracking in Videogame Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hermano Tavares, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gaming Naltrexone Eye Tracking
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Gaming Disorder
Keywords: Videogame disorder; Gaming disorder; eye tracking; naltrexone; problematic videogame users
MeSH Terms: interventions — Naltrexone; Bulk Drugs; Eye-Tracking Technology

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to two groups:
  1. Naltrexone and brief psychoeducational intervention
  2. Placebo and brief psychoeducational intervention This will be double-blind controlled study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone (Experimental): A 12 week Naltrexone flexible dose administration plus 4 sessions of a psychoeducational intervention and 4 eye-tracking sessions
  Interventions: Drug: Naltrexone; Behavioral: Psychoeducational; Device: Eye-tracking
- Placebo (Placebo Comparator): A 12 week placebo matching tablets plus 4 sessions of a psychoeducational intervention and 4 eye-tracking sessions
  Interventions: Drug: Placebo; Behavioral: Psychoeducational; Device: Eye-tracking

INTERVENTIONS:
Drug: Naltrexone — Patients will receive daily doses of Naltrexone, starting at 50mg and increasing 25mg per week until reaching 200mg or the maximum tolerated by the patient
  Other Names: Active drug
  Arms: Naltrexone
Drug: Placebo — Patients will receive daily doses placebo matching tablets for the 12 weeks of the study. Throughout this period, possible adverse effects will be monitored weekly.
  Other Names: Inactive drug
  Arms: Placebo
Behavioral: Psychoeducational — Participants will also attend to 4 sessions of psychoeducational intervention in weeks 2, 4, 6, and 8
Device: Eye-tracking — The attentional bias of the participants will be assessed using the Eye-tracking device in 4 moments throughout the study:
  * Before taking the first dose of naltrexone or placebo.
  * One hour after taking the first dose of naltrexone or placebo.
  * One week after continuous and daily use of naltrexone or placebo.
  * At the end of the intervention, after 12 weeks of continuous and daily use of naltrexone or placebo.
  Other Names: Tobii eye-tracker

SUMMARY:
It is a double blind controlled study to test the hypothesis that it's possible to predict the response to naltrexone in Videogame Disorder with the use of Eye Tracking device, during a period of 12 weeks

DETAILED DESCRIPTION:
This will be a double blind controlled study in which the investigators will select a specific sample of individuals diagnosed with a video game disorder representing a picture of genuine dependence on this technology. The sample will be submitted to the use of naltrexone over a period of 12 weeks and it wiil be assessed whether there was a response to this intervention and whether that response can be predicted through attentional bias analysis using the Eye Tracking device.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be evaluated initially in a clinical interview by a specialized psychiatrist and then by a second interviewer who will use a semi-structured interview to check the DSM-5 criteria for Video Game Disorder (VGD) modeled in the standard format of Schedules for clinical assessment in neuropsychiatry (SCID). Only a specific subgroup of VGD will be included in our sample, which will be called VGDa, a sample that represent a framework of behavioral dependence in essence. Patients in this sample must necessarily have the following symptoms: salience, withdrawal, relapse, conflict, mood modification and fissure. The criteria to delimit this subgroup are listed below:
* Patients diagnosed with Internet Gaming Disorder according to DSM-5
* Patients who have a score of 4 or higher on the following questions on the IGDS9-SF scale (Internet Gaming Disorder Scale 9 - Short Form):

Question 1: Salience assessment. Question 2: Abstinence assessment. Question 4: Relapse assessment. Question 6: Conflict assessment. Question 8: Mood modification assessment.

* Patients with craving according to the adaptation of the Gambling Follow-up Scale (GFS) described below.

An adaptation of the GFS scale, originally used to evaluate patients with Gambling Disorder, was made in order to allow the evaluation of the craving symptom in a patient with VGD. It will only be used the fourth question on this scale as follows.

"4) In the past 4 weeks, how was your desire to play?

1. I felt an irresistible urge to play.
2. I felt a strong desire to play, sometimes resistable, sometimes not.
3. I felt a strong desire to play, but resistable most of the time.
4. I felt a slight desire to play.
5. I didn't feel like playing. " It will considered that the patient has craving if he answers this question by selecting items 1, 2 or 3.

Patients must meet the following criteria before randomization:

* Have read and signed the informed consent form after the nature of the study has been fully explained and before carrying out any procedures related to the study;
* Age between 18 and 60 years old, inclusive;
* Female patients must be:

  1. In post-menopause for at least one year, or;
  2. Being surgically incapable of becoming pregnant (undergoing bilateral hysterectomy or oophorectomy or tubal ligation or otherwise being unable to become pregnant), or;
  3. Be practicing an acceptable method of birth control (defined as: hormonal contraceptives, spermicide plus barrier, a single vasectomized partner and / or intrauterine device).
  4. If a patient with the potential to become pregnant is practicing an acceptable method of birth control (as mentioned above), she must have a negative urine pregnancy test at the enrollment stage, as well as, at baseline, before receiving the study drug.

Exclusion Criteria:

* - Established contraindication to naltrexone (opioid dependence, in the process of opioid withdrawal or current use of opioid analgesics) or hypersensitivity to naltrexone;
* Exposure to any other drug or experimental device in the 30 days prior to inclusion, except for occasional use of benzodiazepines;
* Pregnancy, breastfeeding or patients who intend to become pregnant during the study;
* Evidence of renal failure, defined as serum creatinine levels> 133 mmol / L in men and> 124 mmol / L in women, which correspond to> 1.51 mg / dl and> 1.41 mg / dl, respectively on Week 1 of inclusion;
* Evidence of clinically significant liver failure (defined as AST or ALT> 2 times the upper limit of normal) in Week 1 of inclusion;
* Significant cardiovascular disease, including a history of myocardial infarction in the last 5 years, stroke, clinically significant heart valve disease, unstable angina, clinically abnormal ECG, arrhythmia or congestive heart failure, determining functional class III or IV (NYHA, 1964);
* Uncontrolled hypertension (defined as a diastolic blood pressure of 100 mm / Hg and / or a systolic blood pressure of 180 mm / Hg with or without medication). Hypertensive patients receiving medication should be receiving the same dose of the same antihypertensive medication for at least two months;
* Evidence of uncontrolled thyroid disorders, including hyper or hypothyroidism or abnormal TSH level. Patients who are known to have thyroid hormone replacement need to have had a stable dose for at least three months prior to inclusion and a normal TSH level upon inclusion
* History or current comorbidity with bipolar affective disorder, obsessive compulsive disorder, psychotic disorder, schizophrenia or severe depression, additionally verified through the Patient Health Questionnaire 9 (PQH-9> 19), current suicide risk, or any other neuropsychiatric condition in severe cognitive impairment;
* Current or previous history (in the previous two years) of abuse / dependence on alcohol or other psychoactive substance (except nicotine);
* If at any moment the clinician responsible for the patient identifies suicidal ideation with risk of self-harm, or death;
* Clinically significant hematological or immunological disorder;
* Patients currently receiving psychotropic medications, except for the episodic use of benzodiazepines;
* Illiteracy, or any other condition that prevents the reading and understanding of the research instruments;
* Do not have a telephone line available for remote monitoring;
* Living alone, or not being able to present a family member capable of providing collateral information on gaming behavior;
* To be followed up in another therapeutic program.

The Mini International Neuropsychiatric Interview (MINI) will be used to verify the psychiatric exclusion diagnoses. This is a structured diagnostic interview, with quick application - approximately 45 minutes - compatible with the DSM-IV criteria. Its objective is the verification and standardization of the main Psychiatric Disorders of Axis 1 of DSM IV. It is performed by clinicians after rapid training (1 to 3 hours). The translated and adapted Brazilian version showed globally satisfactory reliability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adpated Internet Gaming Disorder Scale-Short Form (IGDS9-SF) | 12 Weeks.
  IGDS9-SF is 9 items scale in which the patient must answer how often he performs a certain behavior in the last 12 months, the score ranges from 9 to 45, patients with 21 points or more are diagnosed with Video Game Disorder according to the Brazilian validation carried out in 2020.
  As the IGDS9-SF is a diagnostic scale, the adaptations described below were necessary to use it to assess the response to the intervention:
  * Reduction of the time interval to which the scale questions refer, from 12 months to the last 12 weeks.
  * Adaptation of the text of each item in order to reflect the interaction with the video game and its repercussions in the last 12 weeks.
  To validate these changes, the investigators will perform a cross-validation with the Gambling Follow-up Scale adapted for video games described in the next item.
  The application of the adapted IGDS9-SF will occur at the beginning of the follow-up, before the intervention, and at the end of the intervention.
Gambling Follow-Up Scale adapted to Videogames (Gaming Follow-up Scale) | 12 Weeks
  The Gambling Follow-up Scale (GFS) is a self-administered scale of ten items for assessing pathological gamblers throughout treatment. For the use of GFS in this study, the third and fifth questions were excluded, which assessed the financial impact due to gambling, a rare situation in patients with Video Game Disorder (VGD). The eighth question were adapted in order to assess whether the patient had time to dedicate himself to his basic needs, a question that is more congruent to the psychopathology of VGD. And finally, the text of all the questions were adapted by exchanging the word gambling for video games.
  This adapted scale will be applied at the beginning of patient follow-up, before the intervention, being reapplied in 4 weeks and at the end of the intervention in the 12th week.
  To validate this adaptation, the investigators will do a cross-validation with the adapted IGDS9-SF scale described in the previous item.

SECONDARY OUTCOMES:
Gaming Timeline Follow-Back Method (TFB) | 12 weeks
  TFB is a retrospective interview technique designed to assess alcohol consumption. It has been used in a similar way to address other impulsive behaviors, for example, gambling. In this study it will be used to assess the patient's dedication to the video game.
  With this technique, the interviewer obtains information about the days and the amount of resources and time invested in the behavior. Initially, the interviewer identifies relevant dates for the patient in this period and uses them as markers that facilitate the recall of information. It helps and encourages the patient to recall, retrospectively, information about episodes of excessive gaming and write them down on a calendar sheet. Thus, a diary of the activity is obtained in the desired period.
Short Impulsive Behavior Scale (UPPS-P) | 12 weeks
  The Short UPPS-P, like the original UPPS-P, is a Likert scale with 4 possible answers for each item (from Strongly Agree to Strongly Disagree). This scale takes the form of self-report and has 20 items, which then produce scores for the five factors of impulsivity. Each factor ranges from 4 to 16, being the lower values indicative of dysfunctionality. This brief version was successfully validated in English, successfully replicating the internal consistency and the correlations between the factors of the original scale with the benefit of saving about 66% of the time required for application.
Social Adjustment Scale self-report version (SAS) | 12 weeks
  SAS is considered the most carefully developed social adjustment scale, showing the highest levels of reliability and validity. It is widely used and cited in the scientific literature, being useful to assess social adjustment in a wide variety of populations, both clinical and non-clinical. SAS allows an assessment of social adjustment in seven areas: work outside the home, work at home, studies, social life and leisure, relationship with family, spouse, children, home life and financial situation. It consists of 54 questions with 5 possible answers, with higher scores indicating greater impairment. In this study, it will be used to verify the effect of experimental treatment on social adjustment as a secondary outcome.
Global Clinical Scale | 12 weeks
  The Global Clinical Scale will be used to assess global severity, considering the frequency and intensity of symptoms. It is applied by a trained person. Its score varies between 1 (normal, not sick) and 7 (extremely sick). The criterion used for improvement (positive response to treatment) is 1 = improved and 2 = greatly improved.
Rotter's Locus of Control Scale | 12 weeks
  The prediction analysis in this study will be based on individual variation characteristics, more specifically on the internal-external control locus trait, for this the Rotter scale translated and adapted to Brazilian Portuguese will be used. It consists of 29 questions with 2 possible answers, with higher scores indicating External Locus of Control and lower scores indicating Internal Locus of Control
Eye tracking | 12 weeks
  The purpose of this intervention is to carry out assessments of the visual tracking patterns and verify their correlation with the clinical response of the individuals who underwent the intervention.
  The slide shows projected in the test will consist of neutral and video game related images. Each attempt will contain two images (video games and neutrals) and will last for 8 seconds, with 25 attempts in total. Each of the four eye tracking sessions will contain an exclusive slide show (that is, new images each time) and the order of presentation will be random. The dependent variables that will be measured will include: total number of fixations, average length of stay and duration of the first fixation in a video game figure.
Mini International Neuropsychiatric Interview (MINI) | 12 weeks
  Compared with several reference criteria, in different contexts (psychiatric units and primary care centers), this structured diagnostic interview showed psychometric qualities similar to more complex standardized diagnostic interviews and allows a reduction of at least 50% in the evaluation time, with duration 15 to 30 minutes. It will be used in this study to describe and control DSM-IV Axis 1 psychiatric disorders. MINI has a translated and adapted version for Brazil and will be used in this study to control psychiatric comorbidities.
PHQ-9 Patient Health Questionnaire | 12 weeks
  PHQ-9 is one of the most studied psychometric assessment tools for assessing depression in medicine. It is part of a more comprehensive and entirely self-administered test, the PHQ, developed with the aim of screening for frequent mental disorders in the context of primary care such as depression, alcohol use anxiety, somatoform disorders and eating disorders.
  PHQ-9 consists of nine questions, which correspond to the DSM-5's nine diagnostic criteria for depression. Each item receives a score from 0 to 3, indicating the frequency of the presence of symptoms in the last two weeks. The total score ranges from 0 to 27 and represents the sum of the responses of the nine items.
Beck Anxiety Inventory (BAI) | 12 weeks
  The Beck Anxiety Inventory is a self-administered scale composed of 21 questions that measure the intensity of anxiety symptoms in the last week (0 = absent to 3 = severe) through descriptive statements and does not aim at diagnostic aspects. The proposed cut-off note for the Portuguese version, in samples from psychiatric patients, suggests:
  <10 = minimum; 10-19 = light 20-30 = moderate; 31-63 = severe. This scale will be used in this study to control the associated anxious symptoms.
Ugvalg for Kliniske Undersgelser (UKU) scale of side effects | 12 weeks
  The UKU is a detailed scale for assessing drug side effects comprising the following 4 groups of psychic, neurological, autonomic and other side effects. Each item is evaluated on a scale from zero (absent) to 3 (severe). For each item, the causal relationship with the medication in use (unlikely, possible and probable) is marked. There is also an item of global assessment of the interference of side effects on the patient's daily performance (0 = no side effects, 3 = side effects markedly interfering with performance). There is also another item that assesses the consequence of interference: from 0 = no action to 3 = discontinuation of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hermano Tavares, Principal Investigator — Associate
Locations (1):
- Hospital das Clínicas da faculdade de medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Andrade, A. G. D., Bernik, M. A., Brunfentrinker, P., & Negro Júnior, P. J. (1988). Dados de confiabilidade sobre uma entrevista semi-estruturada para avaliaçäo de tratamentos de alcoolistas: escala de severidade de alcoolismo (ESA). Rev. ABP-APAL, 1-4. — https://pesquisa.bvsalud.org/portal/resource/pt/lil-59975
- See also: Dela Coleta MF. Escala multidimensional de locus de controle de Levenson. Arquivos Brasileiros de Psicologia; 39, 79-97. 1987 — http://bibliotecadigital.fgv.br/ojs/index.php/abp/article/view/19592
- See also: Demetrovics, Z., Urbán, R., Nagygyörgy, K., Farkas, J., Zilahy, D., Mervó, B., ... & Harmath, E. (2011). Why do you play? The development of the motives for online gaming questionnaire (MOGQ). Behavior research methods, 43(3), 814-825. — https://link.springer.com/article/10.3758/s13428-011-0091-y
- See also: Field M, Mogg K, Zetteler J, Bradley BP. Attentional biases for alcohol cues in heavy and light social drinkers: the roles of initial orienting and maintained attention. Psychopharmacology (Berl); 176: 88-93. 2004. — https://link.springer.com/article/10.1007/s00213-004-1855-1
- See also: Galetti AM, Tavares H. Development and validation of the Gambling Follow-up Scale, Self-Report version: an outcome measure in the treatment of pathological gambling.Braz J Psychiatry. 39(1):36-44. 2017 — https://www.scielo.br/scielo.php?pid=S1516-44462017000100036&script=sci_arttext
- See also: Garcia, M. S. (2018). Adaptação da escala UPPS-P e sua aplicabilidade na população brasileira. — https://repositorio.ufmg.br/handle/1843/BUOS-B57FEB
- See also: Grant LD, Bowling AC. Gambling attitudes and beliefs predict attentional bias in non-problem gamblers. Journal of gambling studies; 31(4): 1487-1503. 2015. — https://link.springer.com/article/10.1007/s10899-014-9468-z
- See also: Griffiths, Mark. Technological addictions. In: Clinical psychology forum. Division of Clinical Psychology of the British Psychol Soc, 1995. p. 14-14. — https://scholar.google.com.br/scholar?hl=pt-PT&as_sdt=0%2C5&q=Griffiths%2C+Mark.+Technological+addictions.+In%3A+Clinical+psychology+forum.+Division+of+Clinical+Psychology+of+the+British+Psychol+Soc%2C+1995.+p.+14-14.&btnG=
- See also: Hodgins DC. Implications of a brief intervention trial for problem gambling for future outcome research. J Gambl Stud 21:9-13. 2005. — https://link.springer.com/content/pdf/10.1007/s10899-004-1917-7.pdf
- See also: Kim SW, Grant JE. An open naltrexone treatment study in pathological gambling disorder. Int Clin Psychopharmacol; 16(5): 285-9. 2001. — https://journals.lww.com/intclinpsychopharm/fulltext/2001/09000/an_open_naltrexone_treatment_study_in_pathological.6.aspx
- See also: Lahti T, Halme JT, Pankakoski M, et al. Treatment of pathological gambling with naltrexone pharmacotherapy and brief intervention: a pilot study. Psychopharmacol Bull; 43(3): 35-44. 2010. — https://www.ncbi.nlm.nih.gov/pubmed/21150845
- See also: Lole L, Li E, Russell AM et al.. Are sports bettors looking at responsible gambling messages? An eye-tracking study on wagering advertisements. Behav Addict; 1;8(3):499-507. 2019. — https://akjournals.com/view/journals/2006/8/3/article-p499.xml
- See also: McGrath DS, Meitner A, Sears CR. The specificity of attentional biases by type of gambling: An eye-tracking study. PLoS One.;13(1):e0190614. 2018 — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0190614
- See also: Mitchell, J., Tavares, V., Fields, H. et al.. Endogenous Opioid Blockade and Impulsive Responding in Alcoholics and Healthy controls. Neuropsychopharmacol 32, 439-449; 2007. — https://www.nature.com/articles/1301226
- See also: Nestler EJ. From neurobiology to treatment: progress against addiction. Nature Neuroscience; 5: 1076-1079. 2002. — https://www.nature.com/articles/nn945
- See also: Nicoli de Mattos, C., & Tavares, H. (2019). Development and validation of the compulsive-buying follow-up scale: A measure to assess treatment improvements in compulsive buying disorder. Psychiatry Research, 282, 112009-112009. — https://europepmc.org/article/med/30612719
- See also: Şalvarli, Şerife İnci; Griffiths, Mark D. The Association Between Internet Gaming Disorder and Impulsivity: A Systematic Review of Literature. International Journal of Mental Health and Addiction, p. 1-27, 2019. — https://link.springer.com/content/pdf/10.1007/s11469-019-00126-w.pdf
- See also: Santos, Veruska Andrea et al. Treatment of Internet addiction with anxiety disorders: Treatment protocol and preliminary before-after results involving pharmacotherapy and modified cognitive behavioral therapy. — https://www.researchprotocols.org/2016/1/e46/?utm_source=TrendMD&utm_medium=cpc&utm_campaign=JMIR_TrendMD_1
- See also: Sediyama Nogueira, C. Y., Massote Carvalho, A., Gauer, G., Tavares, N., de Miranda Monteiro Santos, R., Ginani, G., ... & Fernandes Malloy-Diniz, L. (2013). Translation and adaptation of impulsive behavior scale (UPPS) to the Brazilian population. — http://search.ebscohost.com/login.aspx?direct=true&profile=ehost&scope=site&authtype=crawler&jrnl=17244935&asa=Y&AN=90478141&h=sZE1F%2BdXEm8Cl8VPk0hNEemPoh%2F4zp9E9ynFj5zseH85%2FfRfwCUuo7mVFHS5STPnVvAa4apfhnnZJGJCyIUGhw%3D%3D&crl=c
- See also: Shao, Rong; WANG, Yunqiang. Effect of Violent Video Games on Adolescent Aggression: Moderated Mediation Effect of Family Environment and Normative Beliefs. Frontiers in psychology, v. 10, p. 384, 2019. — https://www.frontiersin.org/articles/10.3389/fpsyg.2019.00384/full
- See also: Sugaya, Nagisa et al. Bio-psychosocial factors of children and adolescents with internet gaming disorder: a systematic review. BioPsychoSocial medicine, v. 13, n. 1, p. 3, 2019. — https://link.springer.com/article/10.1186/s13030-019-0144-5
- See also: Tavares H, de Brito AM et al..Topiramate Combined with Cognitive Restructuring for theTreatmentof Gambling Disorder: A Two-Center, Randomized, Double-Blind Clinical Trial. J Gambl Stud.;33(1):249-263. 2017. — https://link.springer.com/content/pdf/10.1007/s10899-016-9620-z.pdf
- See also: Van denBrink W. Evidence-based pharmacological treatment of substance use disordersand pathological gambling. Curr. Drug Abuse Rev.; 5(1), 3-31. 2012 — https://www.ingentaconnect.com/content/ben/cdar/2012/00000005/00000001/art00002
- See also: Vitaro F, Hartl AC, et al..Genetica nd environmental influences on gambling and substance use in early adolescence. Behav Genet; 44(4):347-55. 2014. — https://link.springer.com/article/10.1007/s10519-014-9658-6
- See also: Yvonne, H., Yau, M., &Potenza, MD, N. Gambling Disorder and Other Behavioral Addictions: Recognition and Treatment. Harvard Review of Psychiatry; 23, 134-146. 2015. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4458066/